CLINICAL TRIAL: NCT07233044
Title: Effect of Visually-Guided Gait Training on Balance, Mobility and Risk of Falling in Patients With Multiple Sclerosis: A Randomized Controlled Study
Brief Title: Effect of Visually-Guided Gait Training on Balance, Mobility and Risk of Falling in Patients With Multiple Sclerosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Manar El-Sayed Reda Abd El-Fattah, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005505
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visually-guided gait training + Conventional gait training (Experimental): This group will consist of twenty patients, who will receive visually-guided gait training and conventional gait training for 8 weeks.
  Interventions: Other: Visually-guided gait training; Other: Conventional gait training
- Conventional gait training (Active Comparator): This group will consist of twenty patients, who will receive conventional gait training only for 8 weeks.
  Interventions: Other: Conventional gait training

INTERVENTIONS:
Other: Visually-guided gait training — The program runs for eight weeks, with two 60-minute sessions per week, integrating gaze strategy, task-specific mobility, and dual-task cognitive training. Participants first learn systematic visual scanning using saccades and gridline searches. In task-specific training, they perform precision walking-stepping accurately on targets-and obstacle avoidance, navigating a 6 m path with variable pole positions to enhance visual-motor coordination. Finally, dual-task training adds cognitive challenges, such as word generation or backward counting, to improve attention, adaptability, and functional mobility.
  Arms: Visually-guided gait training + Conventional gait training
Other: Conventional gait training — It will be received for eight weeks, twice per week, each session lasting 30 minutes, consisting of standing and walking activities maintaining a stable base of support; static postural control exercises, weight shifting and perturbations exercises, weight-bearing exercises through lower limbs; and adequate weight transfer and forward progression with trunk, limb, and pelvic kinematics consistent with safe walking, walking forward and backward, side-stepping, standing and walking on varied surfaces.

SUMMARY:
The aim of this study is to assess both immediate and long-term effects of visually-guided gait training on balance, mobility, and risk of falling in patients with multiple sclerosis.

DETAILED DESCRIPTION:
Balance and mobility impairments are the most common deficits in people with multiple sclerosis (MS), arising early in the disease course and gradually progressing over time, leading to loss of independence and quality of life. Moreover, static, and dynamic balance deficits in MS patients have been demonstrated to play a major role in patients' perception of walking ability during daily life and in predicting future falls. Given the strong impact of balance impairments on MS patients' disability.

Also, it was reported that the ability to coordinate visual information with movement is normally important to interact with the environment. Indeed, visually guided walking requires the brain to maintain an accurate relationship (or visuomotor mapping) between the perceived stepping location and the motor command necessary to direct the foot to that position on the ground with minimal error. Besides, previous research reported that people with MS, with neuronal transmission impairment or lesions on somatosensory ways, are more dependent on visual compensation for maintain balance. As lesions on somatosensory ways alter postural stability as this fundamental feedback is impaired, making a postural compensation and the visual feedback often more necessary to maintain balance.

To overcome these highly disabling issues, different rehabilitative approaches have been proposed so far in the literature. However, rehabilitation interventions in individuals with MS are limited to aerobic, resistance, and combined aerobic and resistance exercises and instrumental adapted exercise modalities including body-weight-supported treadmill walking or robotic technology. Few studies have addressed the effects of external sensory stimulations (visual, auditory) during gait training on motor performance in patients with multiple sclerosis.

So, visually-guided gait training could be beneficial for improvement of balance and mobility measures and decrease risk of falling for people with MS.

ELIGIBILITY:
Inclusion Criteria:

* Clinically definite MS (relapsing and remitting) patients who are stable for at least three months.
* Expanded Disability Status Scale (EDSS) score of ≤ 4 (fully ambulatory, self-sufficient, and able to stand and walk without any aid or orthosis at least 500 meters) to minimize the impact of motor weakness interfering with their ability to perform the task.
* Normal or corrected to normal vision, wearing eyeglasses.
* The age will range from 20 - 45 years.
* All patients with MS were required to report subjective perceived imbalance or history of falls (in the last year)

Exclusion Criteria:

* Patients with any other neurological deficits or orthopedics abnormalities.
* Patients with secondary musculoskeletal complications such as fractures, contractures, or deformities.
* Patients with vision problems that impaired walking ability.
* Patients with severe cognitive impairment or psychological disorders impaired the ability to follow the procedures of the study.
* Patients with cardiovascular and respiratory diseases.
* Patients with serious unstable medical condition or Patients had an acute exacerbation of MS within last month.
* Pregnant women.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-30 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Dynamic Balance Performance (%): | 8 weeks and follow up after 4 weeks.
  The percentage score representing how accurately the participant maintained the red spot path within the designated frame during the dynamic balance test.
  A higher percentage indicates better balance control and greater stability.
Front Average Deviation | 8 weeks and follow up after 4 weeks
  The mean displacement of the participant's center of pressure (COP) in the forward (anterior) direction.
Back Average Deviation | 8 weeks and follow up after 4 weeks
  The mean displacement of the participant's center of pressure (COP) in the backward (posterior) direction.
Right Average Deviation | 8 weeks and follow up after 4 weeks
  The mean displacement of the participant's center of pressure (COP) in the right (lateral) direction.
Left Average Deviation | 8 weeks and follow up after 4 weeks
  The mean displacement of the participant's center of pressure (COP) in the left (lateral) direction.

SECONDARY OUTCOMES:
The Four-Square Step Test (FSST) | 8 weeks and follow up after 4 weeks
  The Four Square Step Test (FSST) is a valid and reliable tool for assessing mobility in patients with multiple sclerosis (MS). It evaluates self-perceived walking limitations and the ability to quickly change direction and step over obstacles. Using four sticks arranged in a cross, participants step forward, backward, and sideways through each square, then reverse the sequence. The time to complete the task (in seconds) is recorded, with two trials conducted after a practice run; the best time is used. Trials are repeated if balance is lost or an obstacle is touched. Longer completion times (>15 s) indicate greater mobility impairment.
The Ten-Meter Walk Test (10MWT) | 8 weeks and follow up after 4 weeks
  The Ten-Meter Walk Test (10MWT) is a widely recognized, valid, and reliable tool for assessing walking speed in patients with multiple sclerosis (MS). It demonstrates excellent inter- and intra-rater reliability. Participants walk 14 meters, with the middle 10 meters timed to exclude acceleration and deceleration phases. The middle ten meters of a fourteen-meter walkway are timed for 3 trails to calculate average walking speed (m/s). The time taken (in seconds) reflects gait efficiency and mobility performance. As slower walking speed strongly correlates with increased fall risk, the 10MWT also serves as an indirect indicator of fall susceptibility in MS patients.
Arabic version of Falls Efficacy Scale-International (FES-I) | 8 weeks and follow up after 4 weeks
  The arabic version of Falls Efficacy Scale-International (FES-I) is a valid and reliable tool for evaluating fear of falling and fall risk in older adults and individuals with multiple sclerosis (MS). It assesses concern about falling during 16 daily activities performed both indoors and outdoors. Each item is rated on a 4-point Likert scale (1 = not at all concerned to 4 = very concerned), reflecting how worried the individual feels about falling, regardless of actual participation in the activity. The total score ranges from 16 to 64, with higher scores indicating greater fear of falling and reduced confidence in maintaining balance.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Abo Bakr, PhD, Study Chair — Professor, Cairo university; Ibrahim Hamoda, PhD, Study Director — Assistant professor, Kafr Elsheikh univeristy
Locations (1):
- Kafrelsheikh University Hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No